CLINICAL TRIAL: NCT05408910
Title: Rifaximin for Treatment of Bloating in Children and Adults With Cystic Fibrosis
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: new drug formulation by the manufacturer
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Nationwide Children's Hospital (Other); University of Minnesota (Other); University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00086338; MOSHIR21-A0-I (Other: Atrium Health)
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Cystic Fibrosis; Abdominal Pain; Small Bowel Disease
Keywords: Cystic Fibrosis; Cystic Fibrosis in Children; Rifaximin; Bloating; Abdominal distension; Abdominal pain; Small intestinal bacterial overgrowth; Intestinal Dysbiosis; People with Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis; Abdominal Pain | interventions — Rifaximin; Tablets

STUDY DESIGN:
Intervention Model Description: This is a parallel-designed multicenter randomized controlled trial of rifaximin versus placebo done in 100 patients with CF age 12 and up and over 30 kg of weight recruited based on bloating and distension symptoms.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Participants in this arm will receive Rifaximin 550 mg three times daily for 14 days.
  Interventions: Drug: Rifaximin 550 MG Oral Tablet [XIFAXAN]
- Placebo (Placebo Comparator): Participants in this arm will receive placebo three times daily for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin 550 MG Oral Tablet [XIFAXAN] — Participants in this arm will receive Rifaximin 550 mg three times daily for 14 days.
  Other Names: XIFAXAN
  Arms: Treatment
Drug: Placebo — Participants in this arm will receive placebo three times daily for 14 days.
  Arms: Placebo

SUMMARY:
Gastrointestinal symptoms are commonly reported in as much as 65% of people with CF even independent of pancreatic enzyme replacement therapy (PERT) and the most frequent of these symptoms are bloating/distension, flatulence, abdominal pain and bowel habit changes. An alteration in the intestinal microbiome due to intestinal dysmotility, inflammation or other changes including pH changes in the intestine related to CFTR gene mutation may cause intestinal dysbiosis leading to a bacterial overgrowth in the proximal small intestine which may explain some of the findings of distension and bloating in CF.

Our small pilot study aims to investigate use of the only FDA-approved antibiotic, rifaximin for a GI syndrome- IBS, to treat bloating and global GI symptoms in CF patients with bloating and distension. Our goal is to recruit patients >12 years and age/sex matched into rifaximin and placebo arms with total of 100 recruited subjects recruited.

DETAILED DESCRIPTION:
Gastrointestinal symptoms are commonly reported in persons with cystic fibrosis-both adults and pediatrics- and these symptoms cause distress, impact patients quality of life, and can lead to poor nutrition. One of the findings from our largest US study of patient-reported GI symptom outcomes in CF called GALAXY, which enrolled 402 adults and children with CF, was the finding of high rates of patient dissatisfaction with current GI treatments as well as commonly reported symptoms of bloating (48%), fullness (67%) with meals and abdominal distension (50%). This study aims to evaluate if this same-nonsystemically absorbed and noninvasive antibiotic can be used to treat similar commonly reported symptoms in people with CF.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed CF diagnosis who are enrolled in the CFF registry.
2. Mild to severe symptom severity defined as abdominal Distention score ≥ 2 and/or bloating score ≥ 2 on a Likert Scale of 0-6)
3. Patient age ≥12 years and ≥ 30 kilograms (~66.15 lbs)
4. Ability to provide informed consent or presence of legally authorized representative (LAR)
5. Ability to take drug or placebo by mouth (Pill must be intact. May not be opened, crushed, or modified to aid in ingestion)

Exclusion Criteria:

1. Subjects who have previously been allergic to rifaximin or had a hypersensitivity to rifamycin or used rifaximin for any reason within three months (12 weeks) of the study start date
2. Subjects with FEV1 < 40 (as measured within the last 12 months) will be excluded from the study given potential risks in subjects with advanced lung disease
3. Subjects who have received a new antibiotic for treatment of an acute pulmonary infection, or antibiotics for any other infection within 4 weeks prior to randomization or during the study period. Cyclic Antibiotics- Inhaled cyclic antibiotics are allowed at any timepoint. Oral or systemic cyclic antibiotics are exclusionary except for prophylactic antibiotics (e.g., azithromycin) which are allowed. New prophylactic antibiotics cannot be started within 4 weeks of randomization.
4. Subjects with a recent pulmonary exacerbation defined as 4 weeks prior to screening will not be enrolled
5. Subjects who are on probiotics will be asked to discontinue the use of probiotics 14 days prior to randomization as probiotics can alter the gut microbiome and cause bloating
6. Subjects with newly initiated cystic fibrosis transmembrane conductance regulator (CFTR) modulator treatments within one month prior to the study
7. Subjects with new onset of distal intestinal obstruction syndrome (DIOS) or constipation
8. Subjects with advanced liver disease defined by:

   * portal hypertension and/or child Pugh B or C cirrhosis
   * or those with elevated liver enzymes-both AST/ALT > 3 times the upper limit of normal at screening
9. Subjects with bilirubin or alkaline phosphatase elevations > 2 times the upper limit of normal at screening will be excluded as this may be related to CFTR modulator use
10. Women of childbearing potential who are pregnant, trying to become pregnant, breastfeeding, or not using an acceptable method of contraception as described in Section 6.2.
11. Known clostridium difficile colitis. Colonization with c. difficile is not exclusionary.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Rifaximin Treatment Group Improvement of Symptoms | Two weeks
  The primary aim and outcome of our study is to show a significant improvement in individual symptoms of abdominal bloating and/or distension, in PwCF (People with Cystic Fibrosis) treated with rifaximin as compared to placebo

SECONDARY OUTCOMES:
Improved ePROS scores | 42 days
  Our secondary aim and outcome will be based on improvements in the overall ePROS scores and sub-scores for bloating and distension as obtained from GALAXY. These questionnaires will be on a Likert scale ranging from 0-6 where 0 is "Not at all" and 6 is "A very great deal"

CONTACTS AND LOCATIONS:
Overall Officials: Baha Moshiree, MD, Principal Investigator — Wake Forest University Health Sciences

REFERENCES:
- [Background] Furnari M, De Alessandri A, Cresta F, Haupt M, Bassi M, Calvi A, Haupt R, Bodini G, Ahmed I, Bagnasco F, Giannini EG, Casciaro R. The role of small intestinal bacterial overgrowth in cystic fibrosis: a randomized case-controlled clinical trial with rifaximin. J Gastroenterol. 2019 Mar;54(3):261-270. doi: 10.1007/s00535-018-1509-4. Epub 2018 Sep 19. PMID 30232597